CLINICAL TRIAL: NCT04434079
Title: Fluid Balance and Body Weight Changes in Critically Ill Adult Patients
Status: Completed | Type: Observational
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-0486
Record Dates: First submitted 2020-06-05; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Critical Illness; Fluid Overload
Keywords: Fluid Balance; Body Weight Change; Critical Illness
MeSH Terms: conditions — Critical Illness; Edema; Body Weight Changes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Included individuals: Adult patients consecutively admitted to the ICU from June to October 2018 are eligible if expected length of stay is superior to 24 hours and no oral nutritional has been offered.
  Interventions: Other: Regular critical care

INTERVENTIONS:
Other: Regular critical care — Clinical demographic data, daily and cumulative FB (input minus output) with and without insensible fluid losses, and daily and total BW changes are recorded, as well as survival outcome.

SUMMARY:
Positive fluid status has been consistently associated with worse prognosis in critically ill adult patients.However, observational studies showed poor agreement between fluid balance and body weight changes. The objective of the study is to compare the measurements of FB and BW over time and to assess correlation with ICU mortality.

DETAILED DESCRIPTION:
Positive fluid status has been consistently associated with worse prognosis in critically ill adult patients. Daily and cumulative fluid balance (FB) is a routine nursing activity in intensive care unit (ICU). In view of the potential for errors in the calculation of FB totals and the problem of accounting for insensible fluid losses, measurement of body weight (BW) changes is an alternative non-invasive method commonly used for estimating body fluid status. Its accuracy over FB assumes a one kilogram change in BW equates to a one liter gain or loss in body fluid volume. However, observational studies showed poor agreement between those measurements, particularly among individuals staying more than a week in ICU possibly due to muscle and fat loss as well as bone demineralization. The objective of the study is to compare the measurements of FB and BW over time and to assess correlation with ICU mortality.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged >18 years-old admitted to ICU;
* Expected length of ICU stay superior to 24 hours.

Exclusion Criteria:

* Individuals receiving oral diet;
* Actual body weight superior to 227kgs or 501lb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients consecutively admitted to the ICU from June to October 2018 are eligible if expected length of ICU stay is superior to 24 hours and no oral nutritional is being offered.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Correlation between daily fluid balance (difference between fluid input and output during 24 hours) and the change on daily weight | At midnight every 24 hours up to patient's ICU discharge or up to 6 months, whichever comes first.
  Correlation between daily fluid balance and weight change (Bland-Altman agreement test)

SECONDARY OUTCOMES:
Correlation between cumulative fluid balance and total weight change | Last day of each patient's ICU hospitalization, up to 6 months
  Correlation between cumulative fluid balance and total weight change (Bland-Altman)
Discriminative power of fluid balance in predicting ICU mortality | Through study completion, up to 6 months
  Area under ROC curve for fluid balance (L). ICU mortality as reference variable.
Discriminative power of body weight changes in predicting ICU mortality | Through study completion, up to 6 months
  Area under ROC curve for body weight change (kg). ICU mortality as reference variable.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Carolina P Antonio, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil